CLINICAL TRIAL: NCT03528304
Title: Native Women's Wellness: Contingency Management for Tobacco Cessation and Weight Loss
Acronym: NWW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington State University (Other)
Responsible Party: Principal Investigator, Dedra Buchwald, Director, Washington State University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 5U48DP001911-02 (NIH)
Record Dates: First submitted 2016-07-20; First posted 2018-05-17 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Overweight; Obese; Smoking
Keywords: Obesity; Overweight; Current smoker; American Indian/Alaska Native
MeSH Terms: conditions — Overweight; Obesity; Smoking

STUDY DESIGN:
Intervention Model Description: We used a 2x2 factorial design to evaluate contingency management (CM) for weight loss and smoking abstinence among women who were both overweight/obese and current smokers. Participants were accordingly randomized in equal numbers into one of four groups: 1) women receiving CM for weight loss, 2) women receiving CM for smoking abstinence, 3) women receiving CM for both weight loss and smoking abstinence, or 4) a non-contingent control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Smoking arm (Experimental): As part of the CM intervention, women attend visits for smoking and weight loss assessment and are rewarded with prizes for abstaining from smoking.
  Interventions: Behavioral: Contingency management
- Weight loss arm (Experimental): As part of the CM intervention women attend visits for smoking and weight loss assessment and are rewarded with prizes for losing some weight.
  Interventions: Behavioral: Contingency management
- Smoking and weight loss arm (Experimental): As part of the CM intervention, women attend visits for smoking and weight loss assessment and are rewarded with prizes for abstaining from smoking and for losing some weight.
  Interventions: Behavioral: Contingency management
- Control (No Intervention): Women attended clinic visits for smoking status and weight loss assessment.

INTERVENTIONS:
Behavioral: Contingency management — Contingency management (CM) is a behavioral intervention that uses gift cards, prizes, or access to privileges to reinforce specific healthy behaviors and lifestyle changes. CM has been used successfully for a range of addictive behaviors, including cigarette smoking and heroin, cocaine, methamphetamine, and other illicit substance use, as well as for reducing psychiatric problems and HIV risk. CM has great potential for treating smoking and overweight/obesity, as it reinforces both short- and long-term behaviors. This is important because both smoking cessation and weight loss are highly prone to short-term relapse,
  Arms: Smoking and weight loss arm; Smoking arm; Weight loss arm

SUMMARY:
A randomized controlled trial for the efficacy of contingency management to encourage smoking cessation and weight loss.

DETAILED DESCRIPTION:
American Indians and Alaska Native (AI/AN) people experience striking disparities in mortality from cardiovascular disease compared to the general U.S. population. Among women of childbearing age, early detection of chronic diseases can be missed because the type of medical care they seek is typically focused on their reproductive health care needs. Yet, chronic disease risk factors, such as smoking and obesity, are common in this age group and can be treated with evidence-based interventions.

The investigators of this study propose to implement a contingency management (CM) intervention that uses gift cards, and prizes to reinforce smoking cessation and weight loss. CM has been used successfully for a range of addictive behaviors, including cigarette smoking and heroin, cocaine, methamphetamine, and other illicit substance use, as well as for reducing psychiatric problems and HIV risk. CM is understudied in the treatment of obesity, and in AI/AN populations but has great potential for treating smoking and overweight/obesity, as it reinforces both short- and long-term behaviors. This is important because both smoking cessation and weight loss are highly prone to short-term relapse, whereas a longer duration of the desired behaviors is associated with greater success in adopting permanent lifestyle change. The investigators will perform a randomized, controlled trial using a 2x2 factorial design to evaluate a 16-week culturally-tailored CM intervention that promotes cigarette cessation and weight loss among overweight/obese AI/AN women who are current smokers. Participants will be randomized to receive either: 1) CM for smoking abstinence, 2) CM for weight loss, 3) CM for both, or 4) a non-contingent control group that will not receive CM for either behavior. The specific aims are to:

1. Quantify the prevalence of overweight/obesity, smoking, high blood pressure, high cholesterol, Type 2 diabetes and/or elevated fasting blood glucose, and depression and anxiety among women of reproductive age (18-44 years) who are patients at a clinic that primarily serves AI/AN people;
2. Determine if women randomized to CM conditions more often quit or reduce smoking and lose weight compared to those in the control group;
3. Determine if the intervention is disproportionately effective for women receiving CM for both smoking abstinence and weight loss, compared to the single-behavior CM groups or the control group;
4. Quantify group differences in secondary cardiovascular disease risk factors after completing the various CM interventions.

STUDY DESIGN OVERVIEW The CM intervention is 16 weeks long and consists of four groups: 1) CM for smoking abstinence, 2) CM for weight loss, 3) CM for both, or 4) a control group that will not receive CM for either behavior. Participants will be asked to go into the clinic twice a week for 16 weeks during the intervention period, and will be asked to complete a baseline visit at the beginning of the study and three follow-up visits one month apart after the intervention is completed (weeks 20, 24, and 28). In each intervention session the women participants will complete a urine test to determine if they have smoked a cigarette within the past 3-4 days, and will be weighed on a dedicated, standardized scale. Other clinical measurements and self -reported outcomes will be collected as well.

ELIGIBILITY:
Inclusion Criteria:

* 1) female, 2) 18-44 years of age, 3) be of AI/AN heritage, 4) not pregnant, or planning to become pregnant in next 4 months, 5) current daily smoker (self reported), 6) overweight (body mass index = 25.0-29.9 kg/m2) or obese (body mass index ≥ 30 kg/m2), 7) not currently participating in a weight loss program, 8) not interested in using Nicotine Replacement Therapy during the intervention or follow up period, 9) no terminal (e.g., cancer) or debilitating chronic disease (e.g., progressive multiple sclerosis) that would prevent full participation, 10) willing and able to attend 2 study visits per week, 11) willing and able to provide written informed consent.

Exclusion criteria: All other women who do not meet the inclusion criteria.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 125 (Actual)
Dates: Start 2010-09; Primary Completion 2014-09 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Weight Loss | 16 weeks
  Weight loss of 1/2lb to 1lb per week
Smoking Cessation | 16 weeks
  Abstain from smoking

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hartmann-Boyce J, Theodoulou A, Farley A, Hajek P, Lycett D, Jones LL, Kudlek L, Heath L, Hajizadeh A, Schenkels M, Aveyard P. Interventions for preventing weight gain after smoking cessation. Cochrane Database Syst Rev. 2021 Oct 6;10(10):CD006219. doi: 10.1002/14651858.CD006219.pub4. PMID 34611902